CLINICAL TRIAL: NCT01219790
Title: STUDY OF PHASE ID'ACIDE ZOLEDRONIC ASSOCIATED WITH A STRONG DOSE Hypofractionated Radiotherapy in Bone Metastases Vertebral Prostate Adenocarcinoma
Brief Title: ZOLEDRONIC ASSOCIATED With Hight Hypofractionated Radiotherapy Dose in Bone Metastases Vertebral Prostate Adenocarcinoma
Acronym: GEMO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD 10/2-S
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Prostate Adenocarcinoma
Keywords: Patients with painful vertebral metastases with a prostate cancer with an indication of analgesic treatment.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- irradiation + zometa (Experimental)
  Interventions: Radiation: external radiotherapy; Drug: Acide zoledronic

INTERVENTIONS:
Radiation: external radiotherapy — All patients receive a total dose of 27 Gy divided into 3 fractions of 9 Gy performed at least 48 hours apart each, for a treatment to J1, J3 and J5
Drug: Acide zoledronic — The administration of zoledronic acid as defined under the Authorisation on the Market.

SUMMARY:
This study will determine the delayed neurotoxicity (12 months) of a hypofractionated high dose irradiation (3 Gy x 9) associated with zoledronic acid.

The administration of zoledronic acid repeat dosages defined under the Authorisation on the Market.

All patients receive a total dose of 27 Gy divided into 3 fractions of 9 Gy performed at least 48 hours apart each, for a treatment to J1, J3 and J5.

ELIGIBILITY:
Inclusion Criteria:

Adenocarcinoma of the prostate metastatic Age> 18 years3.

* Life expectancy> 12 months;
* Performance Index status <3 PSA ≥ 4 ng / ml Zoledronic acid treatment in progress as recommended by the Authority for the Marketing Creatinine clearance above 30 ml / min Lack of maintenance causing disabling pain not lying down long (30 minutes) No history of radiotherapy to the region to be irradiated Absence of neurological signs compression Distance between the metastasis and spinal cord ≥ 5 mm Absence of metastases unstable metastatic epidural spinal cord compression or may require surgery before radiotherapy

Exclusion Criteria:

* Concomitant treatment with a drug testing, participation in another clinical trial within <30 days
* Presence of central system nervous desease (symptoms or progressive), Patient with a severe neurological disease, current manifestations of peripheral neuropathy> grade 2 NCI-CTC V4 Existence of another severe pulmonary disease, liver or kidney, digestive likely to be exacerbated by treatment,
* Untreated with zoledronic acid
* Treatment with a bisphosphonate other than Zoledronic acid
* Clinically significant hypersensitivity to zoledronic acid, other bisphosphonates or to any excipients in the formulation of Zometa.
* Creatinine clearance below 30 ml / min
* History of another primary cancer (except basal cell skin cancer)
* Or demented patient with altered mental status who can not obtain informed consent. / Persons deprived of liberty or under guardianship
* Pain not resulting in maintaining the prolonged supine position (30 minutes)
* PSA below 4 ng / ml
* History of radiotherapy in localized tumor site
* Distance between the metastasis and spinal cord <5 mm
* Monitoring impossible because of psychological, sociological or because of geographical distance.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2014-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Neurological toxicity was defined as NCI-CTC grade V4.de greater than 2. | 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Paul Papin, Angers
  - Centre Léon Bérard, Lyon
  - Centre René Gauducheau, Saint-Herblain